CLINICAL TRIAL: NCT06930287
Title: Footwear Difference in Sports Use in Runners With Functional Equinus: Observational Study
Brief Title: Footwear Difference in Sports Use in Runners With Functional Equinus
Status: Recruiting | Type: Observational
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, PhD. Physiotherapy, Universidad Católica de Ávila
Other Study IDs: 13/12/2024
Record Dates: First submitted 2025-03-31; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Sport Injury
Keywords: halffoot; sports shoe; daily training; competition

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 300 mg Nimbus shoe
  Interventions: Other: 250 mg Nimbus shoe

INTERVENTIONS:
Other: 250 mg Nimbus shoe — lightweight shoe

SUMMARY:
Observational study on Nimbus shoes for daily training with 8mm drop and designed for heavier than normal weight. Shoe weight is 300g with highly structured buttress and upper with internal heat-sealed midfoot for greater lateral stability. This is a Novablast shoe with a mixed profile for training and competition with 8mm drp and higher midfoot compression range with less lateral containment.

ELIGIBILITY:
Inclusion Criteria:

* patients with functional equine
* regular runners

Exclusion Criteria:

* patients with severe heterometry (more than 1 cm).
* Recent lower limb interventions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: regular runners with functional standing equine
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
functional equine | 5 weeks
  footprints measurement with camera and digital goniometer (measured in degrees).

SECONDARY OUTCOMES:
algometry | 5 weeks
  pressure pain threshold measured with digital algometer (measured in Newtons).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge SAORNIL, PhD., Principal Investigator — Universidad Pontificia de Salamanca
Locations (1):
- Universidad Pontificia de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] MacDonald DRW, Neilly D, Littlechild J, Harrold F, Roberts SC. Acute Achilles tendon rupture: Do cast boots produce adequate equinus when used for functional rehabilitation? Foot (Edinb). 2018 Dec;37:1-4. doi: 10.1016/j.foot.2018.07.004. Epub 2018 Oct 12. PMID 30321852
- [Result] DeHeer PA. Equinus and Lengthening Techniques. Clin Podiatr Med Surg. 2017 Apr;34(2):207-227. doi: 10.1016/j.cpm.2016.10.008. Epub 2017 Jan 19. PMID 28257675
- [Result] Rong K, Ge WT, Li XC, Xu XY. Mid-term Results of Intramuscular Lengthening of Gastrocnemius and/or Soleus to Correct Equinus Deformity in Flatfoot. Foot Ankle Int. 2015 Oct;36(10):1223-8. doi: 10.1177/1071100715588994. Epub 2015 Jun 3. PMID 26041542
- [Result] Rodriguez-Sanz D, Losa-Iglesias ME, Becerro de Bengoa-Vallejo R, Palomo-Lopez P, Beltran-Alacreu H, Calvo-Lobo C, Navarro-Flores E, Lopez-Lopez D. Skin temperature in youth soccer players with functional equinus and non-equinus condition after running. J Eur Acad Dermatol Venereol. 2018 Nov;32(11):2020-2024. doi: 10.1111/jdv.14966. Epub 2018 May 18. PMID 29601106
- [Result] Rodriguez-Sanz D, Losa-Iglesias ME, Lopez-Lopez D, Calvo-Lobo C, Palomo-Lopez P, Becerro-de-Bengoa-Vallejo R. Infrared thermography applied to lower limb muscles in elite soccer players with functional ankle equinus and non-equinus condition. PeerJ. 2017 May 25;5:e3388. doi: 10.7717/peerj.3388. eCollection 2017. PMID 28560116
- [Result] Rodriguez-Sanz D, Losa-Iglesias ME, Becerro-de-Bengoa-Vallejo R, Dorgham HAA, Benito-de-Pedro M, San-Antolin M, Mazoteras-Pardo V, Calvo-Lobo C. Thermography related to electromyography in runners with functional equinus condition after running. Phys Ther Sport. 2019 Nov;40:193-196. doi: 10.1016/j.ptsp.2019.09.007. Epub 2019 Sep 25. PMID 31590122